CLINICAL TRIAL: NCT00477841
Title: Self-Expandable Esophageal Radiation Stent:a Randomized Controlled Trial in Patients With Advanced Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southeast University, China (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 320106196208052017
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2007-05

CONDITIONS: Esophageal Cancer
Keywords: esophageal Cancer; Dysphagia; Stent; interstitial brachytherapy
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Esophageal stent placement
Procedure: dysphagia scores
Procedure: complications of therapy
Procedure: survival time of therapy

SUMMARY:
To determine the response to treatment with a novel esophageal stent loaded with 125I seeds for intraluminal brachytherapy versus a conventional covered stent in patients with advanced esophageal cancer.

DETAILED DESCRIPTION:
Esophageal cancer is common in some areas , ranking as the fourth leading cause of death from cancer in China and sixth worldwide. Although the prognosis of surgical resection for esophageal cancer has been improved, more than 50% of such patients are inoperable and have to undergo palliative treatments because of late stage cancer or metastasis. Dysphagia is the predominate symptom of patients with inoperable esophageal cancer. To relieve the dysphagia and improve the quality of life of such patients, brachytherapy has previously been utilized. Recently, stent placement has been widely accepted to be an option for palliation of the symptoms due to the esophageal strictures. However, recurrence of the neoplastic stricture remains a challenge after stent placement. To combine the advantages of the immediate relief of the esophageal dysphagia with the stent placement and radiation therapy with brachytherapy, a novel esophageal stent loaded with 125I seeds has been developed in the authors' institute. The technical feasibility and safety with this new stent has been demonstrated to be adequate in a healthy rabbit model. The current study is designed to demonstrate the preliminary results with this irradiation stent in patients with inoperable esophageal cancer compared to those using a conventional covered stent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary cancer of esophagus,
* Must be dysphagia caused by esophageal cancer,
* Surgically inoperable, but may be metastatic,
* Without esophageal fistulas,
* Must be an inpatient at Zhongda Hospital,
* Life expectancy is over 6 months,

Exclusion Criteria:

* Esophageal fistulas,
* Tracheal compression with symptoms,
* WBC <2000/mm3 and Platelet count <50,000/mm3,
* Concurrent therapies:surgery, chemotherapy,radiotherapy, Traditional Chinese Medicine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Relief of dysphagia measured by dysphagia scores, survival time from the interventional procedure to the last follow-up. | Follow-up in intervals of 1, 3, 6 and 12 months after stent placement

SECONDARY OUTCOMES:
Successful rate of stent placement, Stent-related complications and morbidity, Overall rate of mortality | Follow-up in intervals of 1, 3, 6, and 12 months after stent placement

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD. Ph.D, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Guo JH, Teng GJ, Zhu GY, He SC, Deng G, He J. Self-expandable stent loaded with 125I seeds: feasibility and safety in a rabbit model. Eur J Radiol. 2007 Feb;61(2):356-61. doi: 10.1016/j.ejrad.2006.10.003. Epub 2006 Nov 7. PMID 17085003